CLINICAL TRIAL: NCT01320293
Title: Effect of Immunomodulatory Therapy With Adalimumab on Endothelial Function in Patients With Moderate to Severe Psoriasis
Brief Title: Cardiovascular Effects in Psoriasis Patients Treated With Adalimumab.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Aida Lugo-Somolinos, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABBO-0001
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis
Keywords: Moderate to Severe Chronic plaque type psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 40mg (Experimental): Adalimumab 40 MG/0.8 ML Subcutaneous Solution [HUMIRA] Dose administered every other week for 6 months
  Interventions: Drug: Adalimumab 40 MG/0.8 ML Subcutaneous Solution [HUMIRA]

INTERVENTIONS:
Drug: Adalimumab 40 MG/0.8 ML Subcutaneous Solution [HUMIRA] — 40mg subcutaneously, every other week for 6 months
  Other Names: Humira

SUMMARY:
Severe psoriasis has been demonstrated to be associated with decreased endothelial function and an increase risk of future coronary events. Although systemic therapy with immunomodulatory agents has been shown to improve psoriatic symptoms, its effects on systemic inflammation and endothelial function are unknown.

In this study we want to assess the cardiovascular risks factors, endothelial dysfunction and inflammatory markers before and after treatment of moderate to severe psoriasis with an FDA-approved biologic agent, adalimumab (Humira).

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be male or female and age 18-55 years at time of consent.
* Must be able to adhere to the study visit schedule and other protocol requirements
* Have chronic plaque psoriasis for more than 6 months with a PASI score of 12 or greater at Baseline.
* Females of childbearing potential (FCBP)‡ must have a negative urine pregnancy test at screening (Visit 1).
* Negative PPD at Screening or 3 months earlier.
* Have not used any biologic treatment for psoriasis in the past 12 months.

Exclusion Criteria:

* Inability to provide voluntary consent
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant, trying to become pregnant or breastfeeding
* Prior diagnosis of coronary artery disease (CAD) or heart disease.
* Systemic fungal infection
* History of past or active mycobacterial infection with any species (including Mycobacterium tuberculosis). Latent Mycobacterium tuberculosis infection as indicated by a positive (more than 15mm induration)Purified Protein Derivative [PPD] skin test. Subjects with a positive PPD skin test and documented completion of treatment for latent TB are eligible. Subjects with a positive PPD skin test and not treated or no documentation of completion of treatment are ineligible.
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
* Clinically significant abnormality on the chest x-ray (CXR) at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer)
* History of Human Immunodeficiency Virus (HIV) infection or Hepatitis C
* Positive Hepatitis B Surface antigen at screening
* Malignancy or history of malignancy (except for treated [ie, cured] basal-cell skin carcinomas > 3 years prior to screening)
* History of any demyelinating disorder such as multiple sclerosis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Lugo-Somolinos, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Dermatology Clinical Trials Unit, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share data

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: active
  Adalimumab: 40mg subcutaneously, every other week for 6 months
Period: Overall Study
Arm/Group | Adalimumab
Started | 18
Completed | 16
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [19 to 52]
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Endothelial Function Compared to Baseline.
Description: Percentage change in endothelial function between baseline visit and end of treatment, 6 months. Endothelial function was measured by percent change in brachial artery diameter after flow mediated dilation (FMD%).
Time Frame: 6 months
Population: 17 of 18 participants completed these assessments at both time points due to one of them having an adverse event that required treatment and therefore end of treatment assessments could not be performed.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 17
percent change | -1.414 [-1.86 to -0.97]
Statistical Analysis 1: Comparison: Adalimumab; Null hypothesis: Percent change in endothelial function from baseline visit to end of treatment/month 6 will be zero change. (percent change=0); Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Changes in IL-6 Profile Compared to Baseline
Description: IL6 average concentration in pg/ml at Baseline compared to end of treatment, 6 months.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Adalimumab
Number analyzed (Participants) | 17
pg/ml | -0.92 [-0.93 to -0.91]
Statistical Analysis 1: Comparison: Adalimumab; Null hypothesis: change in IL-6 levels from baseline visit to end of treatment/month 6 will be zero change. (percent change=0); Test type: Superiority or Other; p < 0.05, t-test, 1 sided

3. Secondary Outcome: Changes in Adiponectin Profile Compared to Baseline
Description: Adiponectin concentration in pg/ml measured at Baseline and end of treatment, 6 months.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Adalimumab
Number analyzed (Participants) | 17
pg/ml | 6.125 [-9.24 to 21.49]
Statistical Analysis 1: Comparison: Adalimumab; Null hypothesis: change in adiponectin levels from baseline visit to end of treatment/month 6 will be zero change. (percent change=0); Test type: Superiority or Other; p = 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Duration of study- 6 months
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=18)
allergic drug reaction (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=18)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
heartburn (Gastrointestinal disorders) | 1 (1)
elbow strain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Smaller number of subjects analyzed due to low enrollment. Technical problems with Elisa measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days